CLINICAL TRIAL: NCT04925050
Title: A Phase I/IB, First-Time-in-Human, Single Centre, Double-Blind, Randomized, Placebo-controlled, Dose Escalating Study of the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of VB0004 Administered Orally to Healthy Volunteers; and to Patients With Mild to Moderate Hypertension With Low Cardiovascular Risk.
Brief Title: First-in-Human Study of VB0004 in Healthy Subjects and to Patients With Mild to Moderate Hypertension With Low Cardiovascular Risk
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB004-001
Record Dates: First submitted 2021-05-21; First posted 2021-06-14 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug VB0004 (Active Comparator): Experimental, Single Ascending dose , Multiple Ascending dose in healthy subjects and naive patients with mild or moderate hypertension with low cardiovascular risk
  Interventions: Drug: VB0004
- Placebo (Placebo Comparator): Matching Placebo for VB0004
  Interventions: Other: Matching Placebo for VB0004

INTERVENTIONS:
Drug: VB0004 — Each study part (A,B and C) will be completed sequentially or with partial overlapping. Safety and PK data through at least day 8 from a subsequent cohort will be reviewed by the SMC prior to dosing the fed period of FE cohort. Safety data will be assessed by SMC after completing each cohorts in MAD healthy volunteers and MAD mild Hypertension patients.
  Arms: Drug VB0004
Other: Matching Placebo for VB0004 — Matching Placebo
  Arms: Placebo

SUMMARY:
This will be a single center, Phase I/IB, randomized, double-blind, placebo-controlled, sequential SAD/MAD/FE study, with a patients arm.

The study will be divided into three parts:

Part A: SAD cohorts, with FE evaluation Part B: MAD cohorts with healthy volunteers Part C: MAD cohorts including naïve patients with mild to moderate hypertension and low cardiovascular risk The three parts will be completed sequentially or with partial overlapping.

DETAILED DESCRIPTION:
Part A - SAD Cohorts 1 to 5:

Part 1 will consist of up to 5 cohorts (1 cohort per dose level). Each cohort will include 8 subjects (6 subjects receiving the active study drug and 2 subjects receiving matching placebo), for a total of 40 subjects. Efforts will be made to have gender-balanced cohorts. A staggered dosing schedule will be used for dosing of each cohort and will include 2 sentinel subjects (1 active and 1 placebo) dosed initially, and the remaining 6 subjects dosed at least 24 hours later. Following completion of each dose level, a Safety Monitoring Committee (SMC) will review the safety and tolerability data, as well as available PK data up to the Follow-Up Visit (Day 8), for at least 6 subjects in the respective cohort, in order to make decisions whether to escalate to the next dose level, decrease the next dose level, repeat a dose level, or to not evaluate any additional dose. The FE study will be conducted with 2 cohorts of 8 healthy participants from the SAD study. Subjects from FE Cohort 3 and, if needed, Cohort 4 will receive the study drug under both fasting (in a first period) and fed conditions (in a second period). There will be a washout period of at least 14 days between dosing of the fasting and the fed periods. Safety, tolerability, and PK data through at least to the Follow-Up Visit (Day 8), from a subsequent cohort will be reviewed by the SMC prior to dosing the fed period of FE Cohort. Therefore, the fed period of a FE Cohort could be dosed in parallel of the SAD Cohort receiving two doses higher. The planned SAD dose range is anticipated to be from 2 mg to 300 mg.

Part B - MAD Cohorts 6 to 8 (Healthy Volunteers):

Part B will consist of 3 cohorts (1 cohort per dose level). Each cohort will include 8 subjects (6 subjects receiving the study drug and 2 subjects receiving matching placebo daily for 14 consecutive days), for a total of 24 subjects. Efforts will be made to have gender-balanced cohorts. Part B can be initiated only following review of the safety, tolerability, and PK data following dosing of the SAD Cohort 3 or 4. A staggered dosing schedule might be used for the first dose level, including 2 sentinel subjects (1 active and 1 placebo) initiating dosing first and the remaining 6 subjects initiating dosing at least 24 hours later. Following completion of each dose level, a SMC will review the safety and tolerability data, as well as available PK data for at least 6 subjects in the respective cohort, in order to make decisions whether to escalate to the next dose level, decrease the next dose level, repeat a dose level, or to not evaluate any additional dose. The planned MAD dose range is anticipated to be from 10 mg to 100 mg administered q.d. for 14 consecutive days.

Part C - MAD Cohorts 9 and 10 (Patients with mild to moderate hypertension): Part C will consist of 2 cohorts (1 cohort per dose level). Each cohort will include a maximum of 8 patients with mild to moderate hypertension with low cardiovascular risk (6 subjects receiving the study drug and 2 subjects receiving matching placebo daily for 28 consecutive days), for a total of 16 patients. The doses of VB0004 administered will be determined by the SAD and MAD PK data. Following completion of Cohort 9, a SMC will review the safety and tolerability data, as well as available PK data for at least 6 subjects in the respective cohort, in order to make decisions whether to escalate to the next dose level, decrease the next dose level, repeat a dose level, or to not evaluate any additional dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker (no use of tobacco or nicotine products within 1 month prior to screening), ≥18 and ≤55 years of age, with BMI >18.0 and <32.0 kg/m2.
* Male subjects who are not vasectomized for at least 6 months, and who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from (the first) study drug administration and for 90 days after (the last) study drug administration:

  1. simultaneous use of a male condom and, for the female partner, oral contraceptives containing combined estrogen and progesterone beginning a least 4 weeks prior to screening, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system (e.g. Mirena), and progestogen-only hormonal contraception associated with inhibition of ovulation, placed at least 4 weeks prior to the first study drug administration.
  2. simultaneous use of a male condom and, for the female partner, nonhormonal intrauterine device (IUD) placed at least 4 weeks prior to the first study drug.

Exclusion Criteria:

* Any laboratory test results deemed clinically significant by the Investigator or positive test for HIV, HBsAg, or HCV.
* Clinically significant ECG abnormalities or vital sign abnormalities (systolic BP lower than 90 or over 140 mmHg (except for hypertensive patients), diastolic BP lower than 40 or over 90 mmHg, HR less than 40 or over 100 bpm, or RR less than 10 or over 22 bpm) at screening.
* Orthostatic hypotension at Screening or Day -1 (Systolic BP falls > 20 mm Hg or Diastolic BP falls > 10 mm Hg on standing)
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 375 mL of beer 3.5%, 100 mL of wine 13.5%, or 30 mL of distilled alcohol 40%]).
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2024-01-23 (Estimated)

PRIMARY OUTCOMES:
The occurrence and severity of treatment related adverse events as defined in CTCAE v4.0 to evaluate the safety and tolerability of VB0004 in healthy volunteers. | Upto Day 21 after each study vaccination
  Adverse events observed during single ascending dose (SAD) and multiple ascending dose (MAD) studies
The occurrence and severity of treatment related adverse events as defined in CTCAE v4.0 which are observed during treatment with repeated doses of VB0004 | Upto Day 35 after each study vaccination
  Patients with mild to moderate hypertension (Blood pressure [BP] 140-15/90-99) will be used to evaluate the safety and tolerability of VB0004.

SECONDARY OUTCOMES:
Calculation of the area under the plasma concentration-time curve for VB0004 to define the pharmacokinetic profile of VB0004 in healthy volunteers. | Up to Day 28
  Both single and multiple doses of VB0004 will be used to define the pharmacokinetic profile of VB0004 from zero time to last measurable concentration
Calculation of the area under the plasma concentration-time curve for VB0004 to define the pharmacokinetic profile of VB0004 in patients with mild to moderate hypertension and low cardiovascular risk. | Up to Day 30
  Both single and multiple doses of VB0004 will be used to define the pharmacokinetic profile of VB0004 from zero time to last measurable concentration
Comparison of the area under the plasma concentration-time curve for VB0004 in both fed and fasted states. | Up to Day 28
  Both the fed and fasted states will be used to define whether food intake affects absorption and/or metabolism VB0004 from zero time to last measurable concentration

OTHER OUTCOMES:
Troponin will be measured in plasma as well as blood pressure in supine and standing positions. | Up to 27 days post dose
  Reductions in one or more of the parameters will indicate the potential efficacy of VB0004 to treat hypertension, cardiac or renal disease
Creatinine will be measured in plasma as well as blood pressure in supine and standing positions. | Up to 27 days post dose
  Reductions in one or more of the parameters will indicate the potential efficacy of VB0004 to treat hypertension, cardiac or renal disease
Cystatin C will be measured in plasma as well as blood pressure in supine and standing positions. | Up to 27 days post dose
  Reductions in one or more of the parameters will indicate the potential efficacy of VB0004 to treat hypertension, cardiac or renal disease

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Nucleus Network Pty Ltd, Victor Harbor, Melbourne
  - Scientia Clinical Research, Randwick, New South Whales
  - Nucleus Network Pty Ltd Geelong Site, Geelong, Victoria

IPD SHARING:
Plan to Share IPD: No